CLINICAL TRIAL: NCT03455686
Title: Single-centre Study Exploring the Utility of Hyperpolarized 129Xe Magnetic Resonance Imaging in Healthy Volunteers and Patients With Lung Disease
Brief Title: Exploring the Utility of Hyperpolarized 129Xe MRI in Healthy Volunteers and Patients With Lung Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Parameswaran Nair, Professor of Medicine, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FIRH_Xe0001
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease; Bronchiectasis; Emphysema; Pulmonary Fibrosis; Bronchopulmonary Dysplasia; Alpha 1-Antitrypsin Deficiency; Sarcoidosis, Pulmonary
Keywords: magnetic resonance imaging; hyperpolarized xenon-129; lung function; lung structure
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Bronchiectasis; Emphysema; Pulmonary Fibrosis; Bronchopulmonary Dysplasia; alpha 1-Antitrypsin Deficiency; Sarcoidosis, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with and without lung disease (Experimental): All enrolled patients will undergo pulmonary function testing, questionnaires, 1H MRI, static ventilation and/or diffusion-weighted hyperpolarized 129Xe MRI and sputum induction at one or more timepoints over five years.
  Interventions: Other: Hyperpolarized 129Xe MRI

INTERVENTIONS:
Other: Hyperpolarized 129Xe MRI — Magnetic resonance imaging (MRI) using inhaled hyperpolarized 129Xe gas is a research approach for the non-invasive visualization and measurement of lung structure and function.

SUMMARY:
This is a single centre exploratory study that aims to apply hyperpolarized xenon-129 (129Xe) magnetic resonance imaging (MRI) methods and measurements in individual patients with and without lung disease to better understand lung structure and function and evaluate response to therapy delivered as a part of clinical care.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the ventilation defect percent (VDP), apparent diffusion coefficient (ADC) and/or the signal-to-noise ratio (SNR) obtained by analysis of hyperpolarized 129Xe MRI at one or more time-points (over time in the absence of therapeutic intervention or following clinically indicated therapy) in healthy volunteers and patients with lung disease including but not limited to: asthma, emphysema, COPD, bronchiectasis, sarcoidosis, pulmonary fibrosis, alpha 1-anti-trypsin deficiency, eosinophilic granulomatosis with polyangiitis and bronchopulmonary dysplasia.

This will be a single centre exploratory study in 10 healthy volunteers with normal lung function and no history of lung disease and 50 patients with a clinical diagnosis of lung disease. There is one study visit required for participation. A subset of participants may be asked to return for up to five additional study visits per year for five years. The purpose of additional study visits is to understand how hyperpolarized 129Xe MRI measurements of lung structure and function change over time in the absence of therapeutic intervention or following clinically indicated therapy.

All subjects will visit St Joseph's Healthcare Hamilton and undergo: vital signs, pulmonary function testing, questionnaires, proton (1H) MRI, static ventilation and/or diffusion-weighted 129Xe MRI, and sputum induction. Up to four doses of hyperpolarized 129Xe will be inhaled during a single study visit.

ELIGIBILITY:
Inclusion Criteria for participants with lung disease:

* Male or female aged 18-85 years with diagnosed lung disease including but not limited to: asthma, emphysema, COPD, bronchiectasis, sarcoidosis, pulmonary fibrosis, alpha 1-anti-trypsin deficiency, eosinophilic granulomatosis with polyangiitis and bronchopulmonary dysplasia.
* Subject understands the study procedures and is willing to participate in the study as indicated by the signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Able to read and/or understand English
* Have a diagnosis of lung disease

Inclusion Criteria for healthy volunteers:

* Subjects male or female aged 18-85 years
* Subject understands the study procedures and is willing to participate in the study as indicated by the signature on the informed consent
* Subject is judged to be in otherwise stable health on the basis of medical history
* Able to read and/or understand English
* No current or previous history of respiratory infection or disease

Exclusion Criteria:

* Age < 18 years or >85 years
* Pregnancy prior to or during study
* In the opinion of the investigator, subject is mentally or legally incapacitated, preventing informed consent from being obtained, or cannot read or understand the written material
* Patient is unable to perform spirometry or plethysmography maneuvers
* Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist/3T Manager)
* In the investigator's opinion, subject suffers from any physical, psychological or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia

Exclusion Criteria for healthy volunteers only:

* Current or previous history of respiratory infection or disease
* Current smoker or ex-smoker with ≥10 pack-year history

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Ventilation Defect Percent (VDP) | 1-5 years
  Whole lung and lobe specific ventilation defect percent (VDP) measured from 129Xe static ventilation magnetic resonance images.
Apparent Diffusion Coefficient (ADC) | 1-5 years
  Whole lung and lobe specific apparent diffusion coefficient (ADC) measured from 129Xe diffusion-weighted magnetic resonance images.

SECONDARY OUTCOMES:
Signal-to-noise ratio (SNR) | 1-5 years
  Signal-to-noise ratio (SNR) measured from 129Xe static ventilation and diffusion-weighted magnetic resonance images.

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute for Respiratory Health, St. Joseph's Healthcare, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirby M, Heydarian M, Svenningsen S, Wheatley A, McCormack DG, Etemad-Rezai R, Parraga G. Hyperpolarized 3He magnetic resonance functional imaging semiautomated segmentation. Acad Radiol. 2012 Feb;19(2):141-52. doi: 10.1016/j.acra.2011.10.007. Epub 2011 Nov 21. PMID 22104288
- [Background] Kirby M, Svenningsen S, Kanhere N, Owrangi A, Wheatley A, Coxson HO, Santyr GE, Paterson NA, McCormack DG, Parraga G. Pulmonary ventilation visualized using hyperpolarized helium-3 and xenon-129 magnetic resonance imaging: differences in COPD and relationship to emphysema. J Appl Physiol (1985). 2013 Mar 15;114(6):707-15. doi: 10.1152/japplphysiol.01206.2012. Epub 2012 Dec 13. PMID 23239874
- [Background] Fain S, Schiebler ML, McCormack DG, Parraga G. Imaging of lung function using hyperpolarized helium-3 magnetic resonance imaging: Review of current and emerging translational methods and applications. J Magn Reson Imaging. 2010 Dec;32(6):1398-408. doi: 10.1002/jmri.22375. PMID 21105144
- [Background] Kruger SJ, Nagle SK, Couch MJ, Ohno Y, Albert M, Fain SB. Functional imaging of the lungs with gas agents. J Magn Reson Imaging. 2016 Feb;43(2):295-315. doi: 10.1002/jmri.25002. Epub 2015 Jul 27. PMID 26218920
- [Background] Shukla Y, Wheatley A, Kirby M, Svenningsen S, Farag A, Santyr GE, Paterson NA, McCormack DG, Parraga G. Hyperpolarized 129Xe magnetic resonance imaging: tolerability in healthy volunteers and subjects with pulmonary disease. Acad Radiol. 2012 Aug;19(8):941-51. doi: 10.1016/j.acra.2012.03.018. Epub 2012 May 15. PMID 22591724
- [Background] Driehuys B, Martinez-Jimenez S, Cleveland ZI, Metz GM, Beaver DM, Nouls JC, Kaushik SS, Firszt R, Willis C, Kelly KT, Wolber J, Kraft M, McAdams HP. Chronic obstructive pulmonary disease: safety and tolerability of hyperpolarized 129Xe MR imaging in healthy volunteers and patients. Radiology. 2012 Jan;262(1):279-89. doi: 10.1148/radiol.11102172. Epub 2011 Nov 4. PMID 22056683
- [Background] Svenningsen S, Kirby M, Starr D, Leary D, Wheatley A, Maksym GN, McCormack DG, Parraga G. Hyperpolarized (3) He and (129) Xe MRI: differences in asthma before bronchodilation. J Magn Reson Imaging. 2013 Dec;38(6):1521-30. doi: 10.1002/jmri.24111. Epub 2013 Apr 15. PMID 23589465
- [Background] Svenningsen S, Eddy RL, Lim HF, Cox PG, Nair P, Parraga G. Sputum Eosinophilia and Magnetic Resonance Imaging Ventilation Heterogeneity in Severe Asthma. Am J Respir Crit Care Med. 2018 Apr 1;197(7):876-884. doi: 10.1164/rccm.201709-1948OC. PMID 29313707
- [Background] Svenningsen S, Nair P, Guo F, McCormack DG, Parraga G. Is ventilation heterogeneity related to asthma control? Eur Respir J. 2016 Aug;48(2):370-9. doi: 10.1183/13993003.00393-2016. Epub 2016 May 12. PMID 27174885
- [Background] Kirby M, Svenningsen S, Owrangi A, Wheatley A, Farag A, Ouriadov A, Santyr GE, Etemad-Rezai R, Coxson HO, McCormack DG, Parraga G. Hyperpolarized 3He and 129Xe MR imaging in healthy volunteers and patients with chronic obstructive pulmonary disease. Radiology. 2012 Nov;265(2):600-10. doi: 10.1148/radiol.12120485. Epub 2012 Sep 5. PMID 22952383